CLINICAL TRIAL: NCT04147377
Title: Effects of Behavioral Interventions Based on Sensory Cues on Freezing of Gait in Parkinson's Disease After Subthalamic Nucleus Stimulation
Brief Title: Effects of Behavioral Interventions Based on Sensory Cues on FOG in PD After STN-DBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, BS Jeon, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1910-104-1071
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Freezing of gait; visual cue; auditory cue; subthalamic nucleus; deep brain stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD with FOG (Experimental): Patients with Parkinson's disease who complain of freezing of gait
  Interventions: Behavioral: behavioral intervention based on sensory cues

INTERVENTIONS:
Behavioral: behavioral intervention based on sensory cues — Patients will receive behavior intervention training that includes how to apply visual and auditory cues to freezing of gait in real clinical practice.

SUMMARY:
The investigators aims to assess the effectiveness of behavioral interventions based on sensory cues on freezing of gait in patients with Parkinson's disease after bilateral subthalamic nucleus deep brain stimulation.

DETAILED DESCRIPTION:
Freezing of gait (FOG) leads to falling and is one of the major determinants of quality of life and prognosis in Parkinson's disease (PD). Previous evidence suggests that subthalamic nucleus deep brain stimulation (STN-DBS) improve off-medication FOG but not on-medication FOG in patients with PD. Furthermore, off-mediation FOG persist or even worsen after STN-DBS in some PD patients.

Although visual and auditory cues are known to improve FOG in research setting, it is unclear whether these cues are effective for FOG in real clinical setting. Most previous studies have used wearable devices to use sensory cues, but such devices are difficult to apply in clinical practice.

Therefore, this study aims to investigate the effectiveness of behavioral interventions based on visual and auditory cues in patients with PD after bilateral STN-DBS. Participants undergo clinical evaluations including the Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), Frontal Assessment Battery (FAB), Unified Parkinson 's Disease Rating Scale (UPDRS), Freezing of Gait-Questionnaire (FOG-Q), and the average number of falling over the last week. Then, participants receive behavior intervention training that includes how to apply visual and auditory cues to freezing of gait in real clinical practice. To investigate the education effect, FOG-Q and the average number of falling over the last week are repetitively assessed at 2-week and 4-week follow-ups using a phone call.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease who are aged 30 years or older
* Patients who underwent bilateral subthalamic nucleus deep brain stimulation
* Patients who complain of freezing of gait

Exclusion Criteria:

* Patients who have already used sensory cues for freezing of gait in clinical practice
* Patients with MMSE scores of 18 or lower
* Patients with Hoehn-Yahr scale 5
* Patients who have neurological symptoms associated with neurological disorders other than Parkinson's disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 4-week f/u in FOG-Q subscore (Q4+Q5+Q6) | baseline, after 4 weeks
  The FOG-Q will be used to determine the efficacy of behavior intervention based on sensory cues.
Change from baseline to 4-week f/u in the number of falling | baseline, after 4 weeks
  We will ask about the average number of falling over the last week at baseline and at 4-week f/u.

SECONDARY OUTCOMES:
Change from baseline to 4-week f/u in FOG-Q total score | baseline, after 4 weeks
  The FOG-Q will be used to determine the efficacy of behavior intervention based on sensory cues.
Change from baseline to 2-week f/u in FOG-Q | baseline, after 2 weeks
  The FOG-Q will be used to determine the efficacy of behavior intervention based on sensory cues.
Change from baseline to 2-week f/u in the number of falling | baseline, after 2 weeks
  We will ask about the average number of falling over the last week at baseline and at 2-week f/u.
Change from baseline to 2-week f/u in FOG-Q subscore (Q4+Q5+Q6) | baseline, after 2 weeks
  The FOG-Q will be used to determine the efficacy of behavior intervention based on sensory cues.

CONTACTS AND LOCATIONS:
Overall Officials: Beomseok Jeon, Professor, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No